CLINICAL TRIAL: NCT02578134
Title: Effectiveness of US-guided Percutaneous Electrolysis (EPE®) Versus Placebo in Individuals With Plantar Fasciosis
Brief Title: US-guided Percutaneous Electrolysis (EPE®) in Plantar Fasciosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Head Division, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URJC 09-2015
Record Dates: First submitted 2015-10-14; First posted 2015-10-16 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Plantar Heel Pain, Plantar Fasciosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- US-guided percutaneous electrolysis (Experimental): Patients will receive one weekly session for 5 weeks for 5 weeks of US-guided percutaneous electrolysis. This intervention consists of the application of a galvanic electrical current with an acupuncture needle in the soft tissue, in this case the plantar fascia insertion. In addition, patients will be asked for conducting a best-evidence low-load exercise programs for the intrinsic foot musculature. The exercise program will be asked to be performed on an individual basis twice every day.
  Interventions: Other: US-guided percutaneous electrolysis
- Sham US-guided percutaneous electrolysis (Sham Comparator): Patients will receive one weekly session for 5 weeks for 5 weeks of sham US-guided percutaneous electrolysis. In this case, the acupuncture needle will be inserted in the soft tissue, in this case the plantar fascia insertion without the application of the galvanic electrical current. In addition, patients will be asked for conducting a best-evidence low-load exercise programs for the intrinsic foot musculature. The exercise program will be asked to be performed on an individual basis twice every day.
  Interventions: Other: Sham US-guided percutaneous electrolysis

INTERVENTIONS:
Other: US-guided percutaneous electrolysis — US-guided percutaneous electrolysis consists of the application of a galvanic electrical current with an acupuncture needle in the soft tissue, in this case the symptomatic insertion of the plantar fascia
  Arms: US-guided percutaneous electrolysis
Other: Sham US-guided percutaneous electrolysis — The acupuncture needle will be inserted into the symptomatic plantar fascia but no galvanic electrical current will be applied, the equipment will be turn off. Patients will be blinded to the application of galvanic electrical current.
  Arms: Sham US-guided percutaneous electrolysis

SUMMARY:
Scientific evidence of conservative management of individuals with plantar fasciosis is sometimes conflicting. There is evidence that regular exercise programs are effective for this pain condition. The inclusion of other therapeutic modalities is still controversial. Some authors have suggested that the use of US-guided percutaneous electrolysis (EPE®) maybe useful for the management of chronic tendinopathies; however, no study has investigated the potential placebo effect of this intervention. The objective of this randomized clinical trial is to determine the effectiveness of US-guided percutaneous electrolysis (EPE®) versus sham US-guided percutaneous electrolysis for the management of patients with plantar fasciosis for pain, function, and disability.

ELIGIBILITY:
Inclusion Criteria:

* insidious onset of sharp pain under the plantar heel surface upon weight bearing after a period of non-weight bearing;
* plantar heel pain which increases in the morning with the first steps after waking up;
* symptoms decreasing with slight levels of activity, such as walking.

Exclusion Criteria:

* prior surgery in the lower extremity;
* diagnosis of fibromyalgia syndrome;
* previous physical therapy interventions for the foot region in the previous 6 months
* lidocaine or other injections in the plantar fascia for the management of pain in the previous 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes in disability before and after the intervention | Baseline, one week after the last session, and 3 months after the last session
  The Foot and Ankle Ability Measure (FAAM) will be used to determine function and disability of the lower extremity induced by plantar heel pain

SECONDARY OUTCOMES:
Changes in pain intensity before and after the intervention | Baseline, one week after the last session, and 3 months after the last session
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of plantar heel pain
Changes in thickness of the plantar fascia | Baseline, one week after the last session, and 3 months after the last session
  An ultrasound (US) assessment of the thickness of the plantar fascia will be conducted to determine changes in fascial tissue thickness

CONTACTS AND LOCATIONS:
Locations (1):
- Cesar Fernandez-de-Las-Peñas, Alcorcón, Madrid, Spain